CLINICAL TRIAL: NCT05534594
Title: Prospective, Single-centre, Feasibility Study to Evaluate the Use of 18F-PSMA PET/CT in Patients With Biochemically Active Medullary Thyroid Cancer
Brief Title: Evaluation of the 18F-PSMA Positron Emission Tomography (PET)/CT in Patients With Medullary Thyroid Cancer
Acronym: MIMETIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202200014
Record Dates: First submitted 2022-08-25; First posted 2022-09-09 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Medullary Thyroid Cancer; Medullary Thyroid Carcinoma; Thyroid Carcinoma, Medullary; Thyroid Cancer, Medullary
Keywords: PSMA PET/CT; 18F-PSMA PET/CT; Fluorine-18 Labeled Prostate Specific Membrane Antigen; Prostate Specific Membrane Antigen; Thyroid Cancer; Medullary Thyroid Cancer; Medullary Thyroid Carcinoma
MeSH Terms: conditions — Carcinoma, Medullary; Thyroid cancer, medullary; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Medullary Thyroid Cancer undergoing 18F-PSMA PET/CT (Experimental): Only 1 arm exists in this study.
  Patients with Medullary Thyroid Cancer undergo a PET/CT after receiving the Fluorine-18 labeled prostate specific membrane antigen (18F-PSMA-1007) tracer intravenously. Each patient will undergo this process one time. Patients will receive 3 MBq/kg (+- 10%) in 8,3 ml (maximum 400 MBq). Waiting time after injection is 60 minutes. Scanning time is approximately 45 minutes.
  Interventions: Drug: 18F-PSMA-1007

INTERVENTIONS:
Drug: 18F-PSMA-1007 — As explained under 'Arms'.
  Other Names: Fluorine-18 labeled prostate specific membrane antigen

SUMMARY:
Rationale: In patients with medullary thyroid cancer (MTC), molecular imaging is used to assess the extent of disease in the primary diagnostic process and follow-up period to determine possible therapeutic options. The currently most used tracer in clinical practice, F-18 labelled fluorodeoxyglucose (18F-FDG), does not accurately detect MTC tumors with an indolent growth rate. A new, complimentary tracer is warranted to detect different subtypes.

Objective: The primary objective is to assess the feasibility of using the F-18 labelled prostate specific membrane antigen (18F-PSMA) PET/CT for (re)staging patients with medullary thyroid cancer. The secondary objective is to compare the ability to detect MTC with the 18F-PSMA PET/CT to that of the 18F-FDG PET/CT.

Study design: Prospective, single-centre, feasibility study.

Study population: Patients (18 years of age or older) with biochemically and cytological/histological confirmed MTC, for whom the indication of an 18F-FDG PET/CT for tumor staging has already been determined on clinical grounds.

Main study parameters/endpoints: The primary outcome of this study is the performance (lesion-based//patient-based sensitivity) of the 18F-PSMA PET to detect MTC lesions in patients with cytologically/histologically confirmed disease. Secondarily, the performance of the 18F-PSMA PET will be compared to the 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histological or cytological proven MTC
* Biochemical evidence of disease activity (elevated/increasing calcitonin and/or CEA)
* Clinical indication for an 18F-FDG PET/CT
* Able to follow instructions to participate in the study
* Able to give informed consent

Exclusion Criteria:

* Patients with prostate cancer or renal cell carcinoma
* Pregnant patients
* Recent neck surgery (<3 months ago)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of 18F-PSMA PET/CT for medullary thyroid cancer. | Up to 2 years
  Patient- and lesion-based sensitivity.

SECONDARY OUTCOMES:
Comparison of the performance of the 18F-PSMA PET/CT to a clinically performed 18F-FDG PET/CT. | Up to 2 years
  Comparison of patient- and lesion-based sensitivity. Comparison of Standardized Uptake Values (SUVs).
Correlation between 18F-PSMA uptake in tumor lesions and serum calcitonin values. | Up to 2 years
  Assess the correlation between 18F-PSMA uptake and serum calcitonin (ng/L) values.
Correlation between 18F-PSMA uptake in tumor lesions and serum carcinoembryonic antigen (CEA) values. | Up to 2 years
  Assess the correlation between 18F-PSMA uptake and serum CEA (ug/L) values.
Correlation between 18F-FDG uptake in tumor lesions and serum calcitonin values. | Up to 2 years
  Assess the correlation between 18F-FDG uptake and serum calcitonin (ng/L) values.
Correlation between 18F-FDG uptake in tumor lesions and serum carcinoembryonic antigen (CEA) values. | Up to 2 years
  Assess the correlation between 18F-FDG uptake and serum CEA (ug/L) values.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No